CLINICAL TRIAL: NCT06221514
Title: Effect Of Core Versus Shoulder Muscles Strengthening Program on Tennis Serve Velocity in Young Adult Tennis Players
Brief Title: Effect of Core Versus on Tennis Serve Velocity in Young Adult Tennis Players
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed ElMelhat, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Core training on TS velocity
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Tennis Elbow
Keywords: tennis; serve velocity; strength; core; shoulder; radar gun
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In this study, double-blinding will be optimized to ensure that the participants are unaware of the study's aim and exact details; in addition, the pre- and post-radar gun assessments will be performed by someone other than the researchers, preferably a tennis coach. Furthermore, shoulder and core training will be performed in the BAU gym under the direction and supervision of coaches and physical therapists; the training program will be given and performed with the coaches before implementing them with the participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core Group (Other): Each session will begin with a 5-10-minute core dynamic warm-up exercise.
  The participants then will perform approximately 30 minutes of core exercises using therapy resistance bands. All players will rest for a few seconds between the exercises. The core exercises will include: bicycle crunches with the band placed around the feet, standing knee tucks with the band placed around the feet (without shoulder rotations and while applying posterior pelvic tilts), flutter kicks with the band placed above the ankles, leg raises with knees flexed and no resistance band, and posterior pelvic tilts from a supine position with hold.
  Lastly, the training session will end with a 5-10-minute cool-down.
  Interventions: Other: Core Strengthening Programs
- Shoulder Group (Other): Each session will begin with a 5-10-minute shoulder dynamic warm-up exercise.
  The participants then will perform approximately 30 minutes of shoulder exercises using therapy resistance bands. All players will rest for a few seconds between the exercises. The shoulder exercises will include: internal and external rotations with the elbow flexed and band wrapped around an object of appropriate height, shoulder abduction to 90˚ with band placed under feet for fixation, shoulder flexion to 90˚ with band placed under feet for fixation, and seated rowing with band held in hands while being placed around the feet were all performed in a sitting position to avoid activation of core muscles.
  Lastly, the training session will end with a 5-10-minute cool-down.
  Interventions: Other: Shoulder Strengthening Programs

INTERVENTIONS:
Other: Core Strengthening Programs — The program will be carried out for 3 weeks, 2 times a week, for approximately 50 minutes.
  Each exercise was performed in 3 sets of 15 repetitions.
  Arms: Core Group
Other: Shoulder Strengthening Programs — The program will be carried out for 3 weeks, 2 times a week, for approximately 50 minutes.
  Each exercise was performed in 3 sets of 15 repetitions.
  Arms: Shoulder Group

SUMMARY:
The goal of this randomized controlled trial is to compare the effect of a 4-week core strengthening program on flat serve velocity in amateur young adult tennis players to a shoulder strengthening program.

Participants will serve the tennis ball four times during the initial and final flat tennis serve assessments. Furthermore, participants will be divided into two groups and given different strengthening programs.

Researchers will compare Group A (shoulder strengthening group) and Group B (core strengthening group) to see if there is any difference between the core and shoulder training programs on the flat serve velocity.

DETAILED DESCRIPTION:
Design:

This study was designed as a double-blinded, randomized controlled trial to investigate the effect of a 4-week core strengthening program versus a shoulder strengthening program on the flat serve velocity in amateur young adult tennis players.

Sample Size:

The sample size was estimated using data from websites that provide information on the Lebanese population, the International Tennis Federation (ITF, 2020), and the Lebanese Tennis Federation (LTF). It is estimated that the age range is 18-25 years. accounts for around 13.84% of the 2,000 tennis players in Lebanon, which equates to 276 players. Of these 276, 64 players (23.19%) were professionals (LTF, 2021), 53 players (25%) were estimated as beginners and the remaining 159 were assumed amateur players. By estimation, 39 players (25%) of the 159 players were excluded as per the exclusion criteria. The population size for the study was determined to be a total of 120 players. Using a scientific sample size calculator software (Qualtrics 2021), the confidence level was set to 90%, and the margin of error was set to 10%. The ideal sample size for this study was calculated and determined to be around 44 ± 10% amateur tennis players. According to this calculation, around 50 amateur tennis players will be recruited for this study.

Participants :

The amateur tennis players will be recruited from multiple tennis academies and online platforms in Beirut, Lebanon through an electronic enrollment form. After collecting all the questionnaires, those that meet the inclusion criteria will be selected, and the participants will be contacted later by email, phone calls, or WhatsApp messages with additional information about the length of the study, the training program, and the number of times per week they expect to be seen.

Players will sign an informed consent sheet provided by the Beirut Arab University (BAU) Institutional Review Board (IRB).

Evaluation:

The initial and final assessments will be performed will be completed in an indoor tennis court to limit the air factor interfering and impacting the serve's velocity after receiving consent from one of the academies and, if necessary, paying rent to use it for 1-2 hours. Following approval, the specific shoulder and core training programs will take place in the BAU gym or at the BAU Physical Therapy Outpatient Clinic under the supervision of the therapists.

Materials

Radar Gun :

Radar will be used to measure the serve speed; it will calculate the time elapsed between the ball's emission and the reception of its reflected echo and the distance traveled by the ball between two points (the ball launch point and a second point) (Tubez et al., 2018). The radar that's held by the assessor will be positioned at least 6 ft behind the player and at a height approximate to the center of the racket head at the point of ball contact.

Resistance Bands Therapy resistance bands will be used for the shoulder and core training resistance exercises (Treiber et al., 1998). For the core exercises, the bands will be placed above the knees, ankles, or around the feet while the participants are performing the exercises in various positions. Additionally, the band will be used for shoulder flexion, abduction, IR, and ER exercises while wrapped around different surfaces.

Statistical Analysis The normal distribution of the data will be checked using the Shapiro-Wilk test. Paired t-tests will be used to compare mean differences between pre-and post-test assessment data for the separate experimental and control groups. One-way ANOVA test will used to compare the pre- and post-assessment means between the groups. The relationship between the independent variables (height, BMI, experience, dominant hand) and dependent variables (pre and post-serve velocity) will be described using Pearson's product-moment correlation coefficients (r). The level of significance for all statistical tests will be set at p < 0.05. All statistical analysis will be conducted through the statistical package for social studies (SPSS).

ELIGIBILITY:
Inclusion Criteria:

1. Tennis playing experience between 1 to 3 yrs.
2. Trains 2-3 times per week for a minimum of 1-2 hours per day
3. Trained in flat serve
4. Right and Left-handed Players
5. Females and males
6. Young adults age ranging from 18-25 years
7. Height ranging from 156-186 cm
8. Body mass index (BMI) of 18.5-24.9 kg/m2.

Exclusion Criteria:

1. Players who underwent specific shoulder or core strength training in the past year
2. Players who had a history of UE injury (dislocation, rupture, fracture, surgery ) that prevents them from playing, and with back or knee pain for at least the past year
3. Players with Cardiovascular diseases or metabolic disorders. (ex: DM)

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Serve Velocity Analysis | Baseline
  1. The flat serve speed will measured in miles per hour using the Bushnell Velocity Speed Radar Gun, which measures the speed of the ball up to 90 feet away (10 to 110 mph) within +/- 1 mph accuracy.
  The therapist will hold the radar at least 6 feet behind the player in the center of the baseline, aligning it with the height approximate to the center of the racket head at the point of ball contact and pointing down the center of the service box (Fernandez-fernandez et al., 2013; Myers et al., 2015).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet M. El Melhat, Phd, Study Director — Cairo University
Locations (1):
- Department of Physical Therapy, Faculty of Health Sciences, Giza, Egypt

REFERENCES:
- [Background] Fernandez-Fernandez J, Ellenbecker T, Sanz-Rivas D, Ulbricht A, Ferrautia A. Effects of a 6-week junior tennis conditioning program on service velocity. J Sports Sci Med. 2013 Jun 1;12(2):232-9. eCollection 2013. PMID 24149801
- [Background] Treiber FA, Lott J, Duncan J, Slavens G, Davis H. Effects of Theraband and lightweight dumbbell training on shoulder rotation torque and serve performance in college tennis players. Am J Sports Med. 1998 Jul-Aug;26(4):510-5. doi: 10.1177/03635465980260040601. PMID 9689369
- [Background] Myers NL, Sciascia AD, Westgate PM, Kibler WB, Uhl TL. Increasing Ball Velocity in the Overhead Athlete: A Meta-analysis of Randomized Controlled Trials. J Strength Cond Res. 2015 Oct;29(10):2964-79. doi: 10.1519/JSC.0000000000000931. PMID 25763521
- See also: Lebanese Tennis Federation — https://ltf.tournamentsoftware.com/ranking/ranking.aspx?rid=195